CLINICAL TRIAL: NCT06487598
Title: Pilot Randomized Controlled Trial to Evaluate add-on Effect of Amalaki (Phyllantus Emblica) and Haridra (Curcuma Longa) Along With Insulin on Glycaemic Control in Patients With Type-I Diabetes Mellitus.
Brief Title: To Evaluate add-on Effect of Nisha-Amalaki Tablets Along With Insulin on Glycemic Control in Type 1 Diabetes Patients (RCTNA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Consultant Pediatrician and Deputy Director, Hirabai Cowasji Jehangir Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JCDC/BHR/24/032
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
Keywords: Type-I diabetes mellitus; Haridra; Amalaki; Prameh
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1-Only insulin treatment for type 1 Diabetes patients (Active Comparator): Arm1:-Insulin treatment- 4 times a day (Basal Bolus insulin) Inj Actrapid from Novo-Nordisk company and Inj Lantus from Sanofi company given as per body weight of patient for 3 months.
  Interventions: Drug: inj insulin to one group; Drug: Inj Insulin with Tab Nisha-Amalaki 500 mg twice a day
- Arm2-Insulin with Nisha-Amalaki tablets (Active Comparator): Arm2:-Insulin treatment- 4 times a day (Basal Bolus insulin) Inj Actrapid from Novo-Nordisk company and Inj Lantus from Sanofi company given as per body weight of patient with Tab Nisha-Amalaki Dhootpapeshwar GMP certified 500 mg twice a day for 3 months.
  Interventions: Drug: inj insulin to one group; Drug: Inj Insulin with Tab Nisha-Amalaki 500 mg twice a day

INTERVENTIONS:
Drug: inj insulin to one group — One group- only inj insulin for 3 months.
  Other Names: Inj Insulin
Drug: Inj Insulin with Tab Nisha-Amalaki 500 mg twice a day — second group- Inj Insulin with Tab Nisha-Dhatri 500 mg twice a day

SUMMARY:
Type-I diabetes mellitus (T1DM) is an autoimmune condition, in which the pancreas reduces/stops insulin production. Patients with T DM have to take insulin injections with every meal and also usually a long-acting preparation. In India, approximately 8.6 lakh people suffer from T1DM, and one in six young patients dies without a diagnosis.

Significant advancements are being made in the field of T1DM research, including stem cell therapy, islet cell transplantation, and immunotherapies, which hold promise for the future. However, so far, there is no known permanent cure for T1DM. Thus, treatment of T1DM aims at maintaining normal blood sugar levels through regular monitoring, insulin therapy, diet, and exercise.

Dietary constituents play an important role in the management of T1DM. Studies have shown that the fruits of Phyllanthus emblica Linn, colloquially known as Indian gooseberry (amla), and/or some of its important constituents (including gallic acid, gallotanin, ellagic acid, and corilagin) possess anti-diabetic actions through their antioxidant and free-radical-scavenging properties. Amla has also been reported to prevent or reduce hyperglycemia, cardiac complications, diabetic nephropathy, neuropathy, cataract genesis, and protein wasting. However, clinical trial data with human subjects are limited and preliminary.

Numerous studies also report that turmeric (Curcuma longa) has antioxidant, anti-inflammatory, and anti-diabetic activities and can lower lipid levels. The hypoglycaemic effect of turmeric may be due to increased peripheral glucose utilization, decreased hepatic glucose synthesis, and/or increased insulin secretion.

In Ayurveda, the combination of turmeric (haridra) and amla (amalaki) is strongly recommended for Prameha (Diabetes mellitus).

ELIGIBILITY:
Inclusion Criteria:

1. K/C/O type-I DM for more than 1 year
2. Age above 10 years, (10-18 years) irrespective of sex, religion, and economic status
3. Parents provide consent and children providing assent for the study

Exclusion Criteria:

1. K/C/O type-I DM for more than 1 year
2. Age above 10 years, (10-18 years) irrespective of sex, religion, and economic status
3. Parents provide consent and children providing assent for the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | 3 months
  Change in glycemic control will be assessed using glycated hemoglobin (HbA1c) by standardized assays.
Change in a insulin dose | 3 months
  Change in an insulin dose will be assessed at baseline and after 3 months of intervention by administering a standardised questionnaire.

SECONDARY OUTCOMES:
Change in urinary parameter. | 3 months
  Change in urinary parameter will be assessed by doing albumin:creatinine ratio(ug/mg)
Change in blood parameter-lipid profile. | 3 months
  Chane in cholesterol(mg/dl), triglycerides(mg/dl),Low density Lipoprotein(mg/dl)
Change in Fat (%) | 3 months
  Change in Body composition by using Bioelectrical Impedance Analysis(BIA)
Change in Body composition. | 3 months
  Change in fat mass ( kg) by using Bioelectrical Impedance Analysis(BIA)

CONTACTS AND LOCATIONS:
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No